CLINICAL TRIAL: NCT05948436
Title: The Impact of Mechanical Methods on the Postpartum Haemorrhage Prophylaxis During Caesarean Section; A Randomized-Controlled Trial
Brief Title: The Impact of Mechanical Methods on the Postpartum Haemorrhage Prophylaxis During Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ipek B. Ozcivit Erkan, MD, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37612
Record Dates: First submitted 2023-07-10; First posted 2023-07-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Hemorrhage; Cesarean Section Complications
Keywords: postpartum hemorrhage; cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamp (Experimental): In these patients, we clamped the uterine artery by Darmklemmen clamp after the delivery of the baby before the delivery of placenta. We released the clamp after the suturing of the uterus is finished.
  Interventions: Procedure: Clamping the uterine artery bilaterally during Cesarean section
- Control (No Intervention): Routine Cesarean section is done.

INTERVENTIONS:
Procedure: Clamping the uterine artery bilaterally during Cesarean section — We clamped the uterine artery by Darmklemmen clamp, which grasps the tissue delicately without damage, after the delivery of the baby before the delivery of placenta. The clamp is released after the suturing of Munro-Kerr incision is finished, before bleeding control. The duration of clamping time is recorded.
  Arms: Clamp

SUMMARY:
The rate of heavy blood loss is higher in Cesarean delivery compared to vaginal deliveries. Since postpartum hemorrhage is a life threatening situation to decrease the maternal mortality and morbidity rates, precautions should be taken. In this study, we aim to decrease the amount of postpartum hemorrhage by clamping the uterine artery after the delivery of the baby during Cesarean delivery.

DETAILED DESCRIPTION:
Obstetrical hemorrhage, is the most common cause of maternal mortality and morbidity that could be prevented. It can appear at early and late stage of delivery and after delivery. It Is defined as loss of more than 500 mL of blood in vaginal deliveries, whereas more than 1L of blood during C-section. The rate of heavy blood loss is higher in Cesarean delivery compared to vaginal deliveries. The incidence of postpartum anemia in Europe is 50% while in developing countries like Turkey it rises up to 50-80%. Since postpartum hemorrhage is a life threatening situation to decrease the maternal mortality and morbidity rates, precautions should be taken. To preserve the hemoglobin concentrations and hemostasis and to optimize the patient's results, evidence-based methods should be performed. Given these circumstances, interventions using pharmacological, mechanical and surgical methods are necessary to minimize the blood loss. Uteroronics are the first line treatment options followed by fundal massage, controlled traction of cord and delivery of placenta, bimanual compression, intrauterine hydrostatic balloon. After these interventions, surgical interventions such as compression sutures, bilateral uterine artery ligation, hysterectomy and pelvic tamponade could be performed. In this study, we aim to decrease the amount of preoperative part of postpartum hemorrhage by clamping the uterine artery by Darmklemmen clamp after the delivery of the baby before the delivery of placenta during Cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women gave birth >37 GW
* singleton pregnancy
* with normal fetal development
* Not emergency C-section

Exclusion Criteria:

* C/sections with indications of plasenta prevue or placenta acrreta spectrum
* with amniotic fluid abnormalities
* multiple pregnancies
* threatened preterm labor
* who have preeclampsia or other type of obstetrical complications
* maternal obesity (BMI>30kg/m2)
* maternal cardiovascular disease, hypertension, coagulation defects, women who use anticoagulants
* patients who underwent Cesarean section during active labor

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
The rate of blood loss | during C-section
  by measuring the suction canister
The rate of blood loss | during C-section
  by weighting the gauze+abdominal compress+under pads used during C-section after subtracting the tare
The rate of blood loss | 24 hours
  by comparing the preoperative and postoperative hemoglobin and hematocrit values

SECONDARY OUTCOMES:
Operation time | during C-section
  minutes
Postoperative complications | postoperative 48 hours
  need for relaparatomy, vascular or organ injury
neonatal outcomes | during C-section
  APGAR scores

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Cepni, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, will ve shared after de identification. The data will be available immediately following publication. No end date. The data will be shared to anyone who wishes to access the data. It could be used for any purpose. Data will be available to anyone who proposes. Proposals should be directed to ipekbetulozcivit@gmail.com, and the link will be provided.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication. No end date.
Access Criteria: The data will be shared to anyone who wishes to access the data.

REFERENCES:
- [Derived] Cepni I, Hamzaoglu Canbolat K, Ozcivit Erkan IB, Sayili U, Yuksel Ozgor B, Ozak E, Mahmudova A, Madazli R, Ocal KP. The Cepni modification: using bilateral vascular clamps during caesarean section for intrapartum hemorrhage, a randomized controlled trial. J Turk Ger Gynecol Assoc. 2025 Jun 10;26(2):73-81. doi: 10.4274/jtgga.galenos.2025.2024-10-4. PMID 40495474